CLINICAL TRIAL: NCT05607836
Title: A Pilot, Prospective, Randomized Trial of IntuBrite Versus Macintosh Direct Laryngoscopy for Paramedic Endotracheal Intubation in Out of Hospital Cardiac Arrest
Brief Title: IntuBrite Versus Macintosh for Endotracheal Intubation in Out of Hospital Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RNN/06/20/KE
Record Dates: First submitted 2022-10-28; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Intubation Complication; Cardiopulmonary Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intu-Brite (Experimental): Use of new laryngoscope - IntuBrite for intubation
  Interventions: Device: IntuBrite intubation
- Macintosh (Active Comparator): Use of standard laryngoscope with Macintosh blade for intubation
  Interventions: Device: Macintosh laryngoscope

INTERVENTIONS:
Device: IntuBrite intubation — Use of new laryngoscope IntuBrite for intubation in patients with cardiopulmonary arrest and during resuscitation
  Arms: Intu-Brite
Device: Macintosh laryngoscope — Use of standard Macintosh blade laryngoscope for intubation in patients with cardiac arrest and requiring cardiopulmonary resuscitation
  Arms: Macintosh

SUMMARY:
a randomized, parallel, non-blinded trial in a single Emergency Mdeical Service in Poland within a group of 34 ground ambulances crews, comparing time and first pass success (FPS) for endotracheal intubation (ETI) in DL using the IntuBrite® (INT) and Macintosh laryngoscope (MCL) during cardiopulmonary resuscitation (CPR). intubations will be performed using INT and MCL based on an intention-to-treat analysis. The FPS time of the ETI attempt will be analysed. First attempt success will be counted.

DETAILED DESCRIPTION:
Investigators designed a prospective observational study to compare INT (IntuBrite®, LLC; Vista, CA, USA) and MCL for ETI performed by paramedics in OHCA without an emergency physician on the scene. The main goal was to determine whether INT is superior to using an MCL laryngoscope during a tracheal intubation attempt in nontraumatic OHCA, in terms of time and effectiveness.

The time of intubation was measured using an electronic stopwatch. Time measurement began when the paramedic held the selected laryngoscope and declared their readiness to perform the procedure.

The effectiveness of the first ETI attempt for instrumental airway management for nontraumatic adult OHCA and end-tidal carbon dioxide monitoring was used to confirm correct device placement in all patients.

The degree difficulty of intubation attempts for all of the patients included in the study. A long-term survival and a cost-effectiveness analysis were not included within this trial.

The investigators will collect case report forms (CRFs) from patients after OHCA within a 40-month period.

The average professional experience of the paramedics in instrumental airway management will be noted (DL and LMA). The primary outcome is the FPS time of the ETI attempt performed by the paramedics.

The success rate on the first intubation attempt will be counted.

ELIGIBILITY:
Inclusion Criteria:

* patients in cardiac arrest , requiring cardiopulmonary resuscitation

Exclusion Criteria:

* suspected difficult intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Intubation time | 1 minute
  Endotracheal intubation from grabbing device to placement of tube in the trachea confirmed by EtCO2

SECONDARY OUTCOMES:
Intubation success | 1 minute
  Endotracheal intubation confirmed with EtCO2
intubation complications | 5 minutes
  intubation complications : esophageal intubation, injuries post intubation

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Gaszynski, Principal Investigator — Medical University of Lodz, Poland
Locations (1):
- Medical University of Lodz, Poland, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kluj P, Fedorczak M, Gaszynski T, Ratajczyk P. A pilot, prospective trial of IntuBrite(R) versus Macintosh direct laryngoscopy for paramedic endotracheal intubation in out of hospital cardiac arrest. BMC Emerg Med. 2023 Jun 23;23(1):70. doi: 10.1186/s12873-023-00845-3. PMID 37349703